CLINICAL TRIAL: NCT00201201
Title: Reducing Adverse Self-Medication Behaviors in Older Adults With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: H02-602; R01HL084208 (NIH)
Record Dates: First submitted 2005-09-16; First posted 2005-09-20 (Estimated); Results first posted 2014-02-03 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2013-12

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
Keywords: Older Adults; Primary Care; Hypertension; Adherence
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension | interventions — Early Intervention, Educational; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Education (Experimental): PEP-NG targeted and tailored education intervention
  Interventions: Other: Education Intervention
- Control (Other): Control, intervention is care as usual.
  Interventions: Other: Control

INTERVENTIONS:
Other: Education Intervention — Adults aged 60 and over with hypertension were randomized to usual care and intervention groups. Both groups entered medication taking behaviors on the PEP-NG and answer questions related to knowledge and self-efficacy regarding adverse self-medication behaviors. The education intervention group received a tailored education program.
  Other Names: Personal Education Program - Next Generation (PEP-NG)
  Arms: Education
Other: Control — Control group receiving care as usual after interfacing with the surveys on the PEP-NG
  Other Names: Control group for PEP-NG
  Arms: Control

SUMMARY:
The purpose of this study is to reduce adverse self-medication practices in older adults with hypertension.

DETAILED DESCRIPTION:
BACKGROUND:

Failure of older adults to take medications properly is estimated to be a factor in more than a quarter of emergency room visits and 10 percent of nursing home admissions, with a total cost of over $25 billion annually. It has been estimated that 10 percent of adverse drug events may be attributed to communication failure between the provider and patient. Lack of adherence to prescription medication protocols and adverse self-medication practices can result in drug interactions that can be fatal. In a health environment that promotes polypharmacy for older adults, a group that is less well able to see, hear, and understand medical information than the general population, a need exists to educate both older adults and their providers about the dangers of adverse drug interactions arising from self-medication.

DESIGN NARRATIVE:

The goal is to reduce adverse self-medication practices in older adults with hypertension. A computer program developed for older adults (Personal Education Program or PEP) will be modified as the next generation PEP, (PEP-NG), to include an interface to allow clients to enter self-medication behavior data independently on a wireless, touch screen tablet computer. Data entered on the PEP-NG will be analyzed via a secure server (ProHealth) and program content tailored to the specific adverse self-medication behaviors will be delivered. Summaries of the reported behaviors with corrective strategies will be printed for both patient and provider so the advanced practice registered nurse (APRN) has a good idea of the client's self-medication practices before beginning the face-to-face interview. Thus, the PEP-NG will make optimal use of the client's waiting time and the APRN's clinical time.

Specific aims are at three levels. 1) To design an interface for the PEP-NG with: a) desirable characteristics for both older adults and primary care providers; and b) minimal user burden. 2) To show that APRNs will increase: a) knowledge concerning potential drug interactions arising from older adults' self-medication practices; b) self-efficacy for teaching older adults about potential drug interactions; c) self-efficacy for communicating with older adults about self-medication; and to d) demonstrate satisfaction using the PEP-NG with clients. 3) To show that older adults using the PEP-NG will: a) increase knowledge concerning potential drug interactions arising from self-medication practices; b) increase self-efficacy as to how to avoid potential drug interactions arising from self-medication practice; c) reduce self-reported adverse behaviors associated with potential drug interactions; 4) improve prescription medication adherence; d) achieve target blood pressure readings; and demonstrate e) satisfaction with the PEP-NG and f) the APRN provider relationship. User-sensitive inclusive design methods will be used to develop and test the patient data interface. After beta-testing the PEP-NG in the primary care laboratory, the PEP-NG will be piloted by 10 APRNs affiliated with ProHealth primary care practices. Repeated Measures Analysis of Variance (RM ANOVA) with one within subjects factor (TIME) will be performed on APRNs' outcome measures at time 0, immediate post-instruction, and 3 and 6 months later. APRNs will each recruit 24 clients (240 total) meeting study criteria. The PEP-NG software will randomly assign each APRN's clients to either control (data collection only) and experimental (data collection plus educational intervention with targeted messages). Client outcome will be assessed at 0, 4, 8, 12, and 52 weeks and analyzed as a mixed ANOVA with NURSE and GROUP as between-subjects factors and TIME as a repeated-measures factor. Healthcare utilization will be compared between the 2 groups after 52 weeks and a cost-benefit analysis conducted.

ELIGIBILITY:
Inclusion Criteria for Older Adults:

* Older adult diagnosed with hypertension
* Health literacy score (REALM) of 44 or greater
* Independent physical and cognitive functioning
* Visual acuity of at least 20/100, with corrective lenses

Exclusion criteria for Older Adults:

* less than age 60
* health literacy score below 44 (6th grade)
* not currently prescribed antihypertensive medication
* visual acuity of less than 20/100 (with corrective lenses, if needed)
* inability to meet independent-living and cognitive-functioning ability.

Inclusion Criteria for APRNs:

* Affiliated with ProHealth Physicians, Inc. practice site in CT and/or
* Affiliated with APRN practice sites in CT

Exclusion Criteria for APRNs:

* Not affiliated with primary care practice sites in CT

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2007-09; Primary Completion 2009-12 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia J. Neafsey, RD, PhD, Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

REFERENCES:
- [Background] Alicea-Planas, J., Neafsey, P.J., & Anderson, E. (2012). Using an e-health intervention to enhance patient visits for hypertension; The nurse practitioner perspective. Journal of Communication in Healthcare, 5(4), 239-249.
- [Background] Lin CA, Neafsey PJ, Anderson E. Advanced practice registered nurse usability testing of a tailored computer-mediated health communication program. Comput Inform Nurs. 2010 Jan-Feb;28(1):32-41. doi: 10.1097/NCN.0b013e3181c0484e. PMID 19940619
- [Background] Neafsey PJ, Anderson E, Coleman C, Lin CA, M'lan CE, Walsh S. Reducing adverse self-medication behaviors in older adults with the Next Generation Personal Education Program (PEP-NG): Design and methodology. Patient Prefer Adherence. 2009 Nov 29;3:323-34. doi: 10.2147/ppa.s7906. PMID 20016796
- [Background] Lin CA, Neafsey PJ, Strickler Z. Usability testing by older adults of a computer-mediated health communication program. J Health Commun. 2009 Mar;14(2):102-18. doi: 10.1080/10810730802659095. PMID 19283536
- [Background] Neafsey PJ, Anderson E, Peabody S, Lin CA, Strickler Z, Vaughn K. Beta testing of a network-based health literacy program tailored for older adults with hypertension. Comput Inform Nurs. 2008 Nov-Dec;26(6):311-9. doi: 10.1097/01.NCN.0000336466.17811.e7. PMID 19047879
- [Result] Neafsey PJ, M'lan CE, Ge M, Walsh SJ, Lin CA, Anderson E. Reducing Adverse Self-Medication Behaviors in Older Adults with Hypertension: Results of an e-health Clinical Efficacy Trial. Ageing Int. 2011 Jun;36(2):159-191. doi: 10.1007/s12126-010-9085-9. Epub 2010 Dec 8. PMID 21654869
- [Result] Anderson EH, Neafsey PJ, Peabody S. Psychometrics of the computer-based Relationships with Health Care Provider Scale in older adults. J Nurs Meas. 2011;19(1):3-16. doi: 10.1891/1061-3749.19.1.3. PMID 21560897
- [Result] Alicea-Planas J, Neafsey PJ, Anderson E. A Qualitative Study of Older Adults and Computer Use for Health Education: "It opens people's eyes". J Commun Healthc. 2011 Apr 1;4(1):38-45. doi: 10.1179/175380611X12950033990179. PMID 23243465
- [Result] Strickler, Z., Lin, C., Rauh, C. & Neafsey, P.J. (2008). Educating older adults to avoid harmful self-medication. Journal of Communication in Healthcare, 1(1), 110-128.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant recruitment brochures and posters with the advanced practice nurses' (APRNs) names/practice contact information were placed in practice waiting and examination rooms. Older adults self-referred for the study by calling the practice and making an appointment with the APRN. Recruitment was rolling during Sept. 2007 - June 2009.
Pre-assignment Details: Exclusion criteria were less than age 60; health literacy score below 44 (6th grade); not currently prescribed antihypertensive medication; visual acuity of less than 20/100 (with corrective lenses, if needed); inability to meet independent-living and cognitive-functioning ability.
Groups:
- Education Intervention: PEP education intervention
  Personal Education Program - Next Generation (PEP-NG) : Adults aged 60 and over with hypertension were randomized to usual care and education (intervention)groups. Both groups entered medication taking behaviors on the PEP-NG and answered questions related to knowledge and self-efficacy regarding adverse self-medication behaviors. The education (intervention) group received a tailored education program generated by the PEP-NG software and reinforced by the APRN.
- Control: Control:
  Adults aged 60 and over with hypertension were randomized to usual care and education (intervention)groups. Both groups entered medication taking behaviors on the PEP-NG and answered questions related to knowledge and self-efficacy regarding adverse self-medication behaviors. The control group met with the APRN after entering their data on the PEP-NG but did not receive a targeted and tailored education intervention.
Period: Overall Study
Arm/Group | Education Intervention | Control
Started | 87 | 73
Completed | 82 | 66
Not Completed | 5 | 7
Not completed — Death | 0 | 2
Not completed — Withdrawal by Subject | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Education Intervention: PEP education intervention
  Personal Education Program - Next Generation (PEP-NG) : Adults aged 60 and over with hypertension were randomized to usual care and education (intervention)groups. Both groups entered medication taking behaviors on the PEP-NG and answered questions related to knowledge and self-efficacy regarding adverse self-medication behaviors. The education (intervention) group received a tailored education program.
- Total: Total of all reporting groups
Arm/Group | Education Intervention | Control | Total
Number analyzed (Participants) | 87 | 73 | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 21 | 47
  >=65 years | 61 | 52 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (9.5) | 69.6 (7.7) | 68.6 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 60 | 125
  Male | 22 | 13 | 35
Region of Enrollment [Number; unit: participants]
  United States | 87 | 73 | 160

OUTCOME MEASURES:

1. Primary Outcome: Behaviors Risk Score
Description: Using a five-point scale from 1, "very unlikely" to 5, "very likely," a five-member expert panel rated a list of adverse self-medication behaviors. The weight of each behavior was the mean of the expert ratings. Adverse self-medication behaviors were identified from questions that address use of medications (in the past month) to treat high blood pressure as well as use of OTC agents and alcohol for common problems that were self-treated with non-prescription agents. Participants were also asked if they drank alcoholic beverages, smoked or used nicotine, or took any vitamin or mineral supplements (including what, when and how frequently each was taken). The Adverse Self-Medication Behavior Risk Score is the sum (range 3 - 60) of the scores for the adverse behaviors identified. The higher the score, the higher the risk is for adverse self-medication behaviors.
Time Frame: Measured at 0, 4, 8, and 12 weeks on visit 1, 2, 3 and 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Education Intervention | Control
Number analyzed (Participants) | 82 | 66
units on a scale
  Visit 1 (0 weeks) | 17.9 (15.4) | 16.6 (15.9)
  Visit 2 (4 weeks) | 16.4 (13.4) | 12.6 (12.6)
  Visit 3 (8 weeks) | 15.9 (12.9) | 14.1 (13.3)
  Visit 4 (12 weeks) | 13.4 (11.2) | 14.2 (13.5)
Statistical Analysis 1: Comparison: Education Intervention vs Control; Repeated measures linear-mixed model ANOVA methodology was employed as each participant was measured on 4 visits and the 4 repeated measures are likely dependent. We used study group (intervention vs. control) and visit as categorical variables and controlled for gender, age, APRN, income, education, computer use. Non-parametric tests (Cochran-Mantel-Haenszel statistic), based on rank scores, controlling for participant code were used for the transformed behavior risk scores within groups; Test type: Superiority or Other; p = 0.035, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel statistic (1,161)=4.44,p=0.035)

2. Primary Outcome: Blood Pressure (BP) Readings: Systolic Blood Pressure
Description: BP measurements were taken by the APRN at each of 4 visits - at the beginning of PEP-NG use on visit 1, and post-PEP-NG use on subsequent visits.
Time Frame: Measured at weeks 0, 4, 8 and 12 on visit 1, 2, 3 and 4
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Education Intervention | Control
Number analyzed (Participants) | 82 | 66
mm Hg
  Visit 1 (0 weeks) | 129.1 (15.5) | 127.4 (13.4)
  Visit 2 (4 weeks) | 128.6 (15.2) | 128.8 (13.3)
  Visit 3 (8 weeks) | 125.8 (13.2) | 128.6 (15.6)
  Visit 4 (12 weeks) | 126.5 (13.5) | 128.5 (13.6)
Statistical Analysis 1: Comparison: Education Intervention vs Control; Repeated measures linear-mixed model ANOVA methodology was employed as each participant was measured on 4 visits and the 4 repeated measures are likely dependent. We used study group (intervention vs. control) and visit as categorical variables and controlled for gender, age, APRN, income, education, computer use; Test type: Superiority or Other; p = .0204, ANOVA

3. Secondary Outcome: Self-efficacy for Avoiding Adverse Self-medication Behaviors
Description: The Self-efficacy scale is a 12-item instrument with statements reflecting patient confidence in selecting appropriate OTC agents and supplements, aside from avoiding adverse effects arising from self-medication behaviors. This scale has 5-point self-report response categories (ranging from 1, "Not Sure" to 5, "Totally Sure"). Responses were summed and divided by the number of items answered, so that the overall score would not be affected by omitted items and was reported based on the original 5-point metric. The higher the score on the instrument, the higher the degree of self-efficacy for avoiding adverse self-medication behaviors.
Time Frame: Measured at 0, 4, 8 and 12 weeks on visit 1, 2, 3 and 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Education Intervention | Control
Number analyzed (Participants) | 82 | 66
units on a scale
  Visit 1 (0 weeks) | 2.5 (0.9) | 2.3 (0.9)
  Visit 2 (4 weeks) | 2.7 (0.9) | 2.4 (0.8)
  Visit 3 (8 weeks) | 3.0 (0.8) | 2.6 (0.8)
  Visit 4 (12 weeks) | 3.3 (0.7) | 2.5 (0.8)
Statistical Analysis 1: Comparison: Education Intervention vs Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = .0001, ANOVA

4. Secondary Outcome: Prescription/Over the Counter (Rx-OTC) Knowledge
Description: The OTC-Rx Knowledge scale has 14 multiple-choice items and the score is the percent of the items with correct response (range: 0-100%; these items test both knowledge and application concerning potential adverse effects of self-medication with OTC agents, supplements, or alcohol in persons with hypertension. The higher the score, the higher the knowledge of the potential adverse effects from self-medication.
Time Frame: Measured at 0, 4, 8, 12 weeks on visits 1, 2, 3 and 4
Measure: Mean (Standard Deviation); unit: percentage of questions correct
Arm/Group | Education Intervention | Control
Number analyzed (Participants) | 82 | 66
percentage of questions correct
  Visit 1 (0 weeks) | 45.2 (16.4) | 45.6 (14.6)
  Visit 2 (4 weeks) | 51.0 (16.5) | 44.8 (17.0)
  Visit 3 (8 weeks) | 57.0 (15.3) | 46.4 (16.5)
  Visit 4 (12 weeks) | 59.4 (16.4) | 45.1 (16.2)
Statistical Analysis 1: Comparison: Education Intervention vs Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0001, ANOVA

5. Secondary Outcome: Satisfaction With the PEP-NG
Description: The PEP-NG user Satisfaction scale is a 14-item instrument - with eight items addressing the ease of program use, program content, and suitability of program content - and another six items addressing the intent to change behavior following program use. Ratings reflected by the 5-point Likert-type scale (ranging from 1, "strongly disagree" to 5, "strongly agree") were summed and divided by the number of items answered to ensure that the overall Satisfaction scale was not affected by omitted items and was cast in the original 5-point metric. The higher the score on the instrument, the higher the degree of satisfaction with the PEP-NG.
Time Frame: Measured at 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Education Intervention | Control
Number analyzed (Participants) | 71 | 64
units on a scale | 4.2 (0.5) | 4.0 (0.4)
Statistical Analysis 1: Comparison: Education Intervention vs Control; Test type: Superiority or Other; p = 0.0431, t-test, 2 sided

6. Secondary Outcome: Satisfaction With the APRN Provider Relationship
Description: The Healthcare Relationships Scale assesses the perceived communication relationship with a provider. The 5-item instrument, based on two qualitative studies addresses patient-provider communication (2 questions), trust, decision-making related to care, and satisfaction with care. The scale was modified for use with older adults by changing the visual analog 10 cm response format to 5-point Likert-type responses with two extremes (e.g., 1:"not at all easy" to 5: "very easy").
Time Frame: Measured at 0, 12 weeks on visit 1 and 4
Population: There 69 participants in the control group and 82 participants in the education intervention group who chose to complete the satisfaction with the APRN provider on visit one and 65 in the control group and 75 in the education intervention group who chose to complete the survey on visit 4.
Measure: Mean (Standard Deviation); unit: units on a scale of 1-5
Arm/Group | Education Intervention | Control
Number analyzed (Participants) | 82 | 69
units on a scale of 1-5
  Satisfaction with APRN Visit 1 (0 weeks) | 4.40 (0.68) | 4.46 (0.83)
  Satisfaction with APRN Visit 4 (12 weeks) | 4.34 (0.60) | 4.42 (0.63)
Statistical Analysis 1: Comparison: Education Intervention vs Control; Analyzed at 0 and 12 weeks; Test type: Superiority or Other; p < .10, t-test, 2 sided

ADVERSE EVENTS:
Groups:
- Education: PEP education intervention
  Personal Education Program - Next Generation (PEP-NG) : Adults aged 60 and over with hypertension will be randomized to usual care and intervention groups. Both groups will enter medication taking behaviors on the PEP-NG and answer questions related to knowledge and self-efficacy regarding adverse self-medication behaviors. The intervention group will receive a tailored education program.
- Control: Control group without education intervention.
Arm/Group | Education | Control
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/73
Other Adverse Events (participants affected / at risk) | 0/87 | 0/73

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No